CLINICAL TRIAL: NCT05043038
Title: Effect of Night Float Call on Sleep and Activity Patterns Among Anesthesia Residents
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexandra Ruan, Clinical Assistant Professor, Stanford University
Other Study IDs: 51495
Record Dates: First submitted 2021-08-24; First posted 2021-09-13 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sleep Disorder, Shift Work; Fatigue; Sleep Disturbance
Keywords: Medical Education; Physician Well-Being; Internship and Residency; Work Schedule Tolerance; Fatigue; physician Burnout; Sleep Disruption
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Fatigue; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia Night Float: The residents will be followed over a three week period - one week prior to night float (baseline), the week of night float, and one week after night float (recovery). Participants will be asked to fill out PROMIS surveys weekly.
- Obstetric Anesthesia Rotation: The residents will be followed and asked to wear the fitbit over a four week period during their rotation. Participants will complete three PROMIS surveys over the four week rotation, and as well as a follow-up PROMIS survey one week after the study period has completed

SUMMARY:
With increasing awareness about physician fatigue and its effect on patient safety, residency programs are increasingly transitioning to a night float call system. In other industries, multiple night shifts in a row can cause a disruption in the circadian rhythm, sleep debt, shift work disorder, that is related to chronic medical conditions such as obesity and cardiovascular disease. We will evaluate the effect of different call structures on resident activity, sleep and self reported measures of wellness using a commercially available Fitbit device.

DETAILED DESCRIPTION:
Participants will be recruited via an email once they are scheduled for a week of night float in the Stanford Main Operating room or on their Obstetric Anesthesia rotation. Potential participants who are taking prescription medications that might affect their alertness during the study period will not be enrolled.

The investigators will quantify the changes in sleep pattern and activity during different call rotations. Self reported aspects of well being including fatigue, physical function, and positive affect will be assessed with NIH PROMIS surveys periodically during the study period. The investigators will use the Fitbit Alta HR data to quantify the change in total amount of sleep, sleep interruption and sleep phase and steps per day. Data will be analyzed only when it is coincident with heart rate data to correct for periods when the device is not used.

Activity will not alter from the participants normal except that they will wear the Fitbit and respond to the NIH PROMIS surveys over the study period.

Data from NIH PROMIS surveys, Fitbit and provided demographic information including age, sex and BMI, and number of previous night float periods previously completed. After association, data will be completely de-identified.

All data will be normalized to the participant's baseline value during the run-in week. The call week and post call week will be analyzed with a time series mixed effects model using R and/or NONMEM (a program for Nonlinear Mixed Effects Modeling). The effects of the above demographic variables will be assessed as potential covariates.

The investigators anticipate that this observational study will be the first of many studies looking at the effects of changing sleep patterns on activity and well-being

ELIGIBILITY:
Inclusion Criteria:

* All residents (PGY2-5) who have been scheduled for either general operating room night float call or obstetric anesthesia rotation

Exclusion Criteria:

* Participants who report taking prescription medications that may effect alertness during the study period will not be enrolled.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit participants who are PGY2-5 and part of the Stanford Hospital Department of Graduate Medical Education, which means they will generally be between 26-36 years of age. We will aim to recruit an equal number of males and females which is reasonable give the demographic distribution of Anesthesia residents. Finally, we aim to have a people with a variety of races and ethnicity involved but this will not be specifically targeted or evaluated due to the limited pool of eligible subjects.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Total Sleep Hours During Night Float | 3 weeks
  The investigators will compare total sleep hours per 24 hour period during a baseline week, a night float week, and a recovery week
Change in Rapid Eye Movement Sleep Hours During Night Float | 3 weeks
  The investigators will compare total Rapid Eye Movement sleep hours per 24 hour period during a baseline week, a night float week, and a recovery week
Change in Daily Steps during Night Float Week | 3 weeks
  The investigators will compare Steps per 24 hour period during a baseline week, a night float week, and a recovery week
Trends and Recovery Time in Total Sleep Hours, Rapid Eye Movement, and Daily Steps during a random night call schedule | 4 weeks
  The investigators will compare change in fitbit sleep and steps data during random call night schedule and recovery after the call night during the obstetric anesthesia rotation
Comparison in sleep and activity patters between a night float call schedule and a random night call schedule | 4 weeks
  The investigators will compare trends in sleep hours, REM sleep, and steps between night float and random call schedule. Time to recovery to baseline sleep patterns will be assessed.

SECONDARY OUTCOMES:
Cohort 1: Change in PROMIS Positive Affect, Sleep Disturbance and Fatigue Scores During Night Float Week | 3 weeks
  Participants will take a survey prior to starting night float, at the end of night float week, and after one recovery week. The questions on the PROMIS survey are answered on a Likert scale and normalized to a scale 1-100 based on national average. The mean value for each survey is 50. A higher score would represent increased level of positive affect.
Cohort 2: Change in PROMIS Positive Affect, Sleep Disturbance, and Fatigue Scores throughout the Obstetric Anesthesia Rotation | 3 weeks
  Participants will take a baseline survey prior to starting the rotation, at the halfway point, at the end of the four weeks, and one week after the conclusion of the study period.
Change in PROMIS Positive Affect, Sleep Disturbance and Fatigue Scores over the study period in a night float versus a random call night system | 4 weeks
  The week to week changes in PROMIS scores between night float and a random call system will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Ruan, MD, Study Director — Stanford University; Pamela Flood, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

REFERENCES:
- [Background] Belayachi J, Benjelloun O, Madani N, Abidi K, Dendane T, Zeggwagh AA, Abouqal R. Self-perceived sleepiness in emergency training physicians: prevalence and relationship with quality of life. J Occup Med Toxicol. 2013 Sep 21;8(1):24. doi: 10.1186/1745-6673-8-24. PMID 24053730
- [Background] Asken MJ, Raham DC. Resident performance and sleep deprivation: a review. J Med Educ. 1983 May;58(5):382-8. doi: 10.1097/00001888-198305000-00003. PMID 6343602
- [Background] Cavallo A, Jaskiewicz J, Ris MD. Impact of night-float rotation on sleep, mood, and alertness: the resident's perception. Chronobiol Int. 2002 Sep;19(5):893-902. doi: 10.1081/cbi-120014106. PMID 12405552
- [Background] Davis MC, Kuhn EN, Agee BS, Oster RA, Markert JM. Implications of transitioning to a resident night float system in neurosurgery: mortality, length of stay, and resident experience. J Neurosurg. 2017 Apr;126(4):1269-1277. doi: 10.3171/2016.5.JNS152585. Epub 2016 Jul 8. PMID 27392266
- [Background] Dunn LK, Kleiman AM, Forkin KT, Bechtel AJ, Collins SR, Potter JF, Kaperak CJ, Tsang S, Huffmyer JL, Nemergut EC. Anesthesiology Resident Night Float Duty Alters Sleep Patterns: An Observational Study. Anesthesiology. 2019 Aug;131(2):401-409. doi: 10.1097/ALN.0000000000002806. PMID 31149926
- [Background] Nizamuddin SL, Nizamuddin J, Latif U, Tung A, Klafta JM, Lee SM, Ku CM, Stahl DL, Lee J, Shahul SS. Be Active and Be Well? A Cross-sectional Survey of US Anesthesia Residents. J Educ Perioper Med. 2020 Apr 1;22(2):E640. doi: 10.46374/volxxii-issue2-nizamuddin. eCollection 2020 Apr-Jun. PMID 32939368
- [Background] Lee HA, Lee HJ, Moon JH, Lee T, Kim MG, In H, Cho CH, Kim L. Comparison of Wearable Activity Tracker with Actigraphy for Sleep Evaluation and Circadian Rest-Activity Rhythm Measurement in Healthy Young Adults. Psychiatry Investig. 2017 Mar;14(2):179-185. doi: 10.4306/pi.2017.14.2.179. Epub 2017 Mar 6. PMID 28326116

DOCUMENTS (1):
  • Informed Consent Form (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT05043038/ICF_001.pdf